CLINICAL TRIAL: NCT00343551
Title: A Nine-week, Randomized, Double-blind, Parallel Group Study to Evaluate the Efficacy and Safety of Aliskiren 300 mg Compared to Irbesartan 300 mg and Ramipril 10 mg in the Setting of a Missed Dose in Patients With Essential Hypertension
Brief Title: Efficacy and Safety of Aliskiren 300mg Compared to Irbesartan 300mg and Ramipril 10 mg in the Setting of a Missed Dose for Patients With Essential Hypertension.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2351
Record Dates: First submitted 2006-06-22; First posted 2006-06-23 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Essential Hypertension
Keywords: Hypertension, ambulatory blood pressure, missed dose, aliskiren
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: Aliskiren

SUMMARY:
The purpose of this study is to investigate the efficacy (blood pressure lowering effect) and safety of aliskiren given to hypertensive patients after a missed dose.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients 18 years of age and older.
* Patients must meet following blood pressure criteria:

At Visit 2 : Office Mean Sitting Diastolic Blood Pressure ≥ 90 mmHg and < 110 mmHg At Visit 3 : Office Mean Sitting Diastolic Blood Pressure ≥ 95 mmHg and < 110 mmHg before application of Ambulatory Blood Pressure Measurement device At Visit 3 : 24-hr Mean Ambulatory Diastolic Blood Pressure ≥ 85 mmHg

* Patient must have an absolute difference of ≤ 10 mmHg in their office Mean Sitting Diastolic Blood Pressure between Visit 2 and 3.
* Male or female patients are eligible. Female patients must be either post-menopausal for at least one year, surgically sterile or using effective contraceptive methods such as oral contraceptives, barrier method with spermicide or an intrauterine device. Reliable contraception should be maintained throughout the study and for 7 days after study drug discontinuation.
* Patients who are eligible and able to participate in the study, and who consent to do so after the purpose and nature of the investigation has been clearly explained to them (written informed consent).

Exclusion Criteria:

* Severe hypertension [Office Mean Sitting Diastolic Blood Pressure ≥ 110 mmHg and/or office mean sitting systolic blood pressure (MSSBP) ≥ 180 mmHg].
* Current diagnosis of heart failure (NYHA Class II-IV).
* History of myocardial infarction, coronary bypass surgery, or any percutaneous coronary intervention (PCI) during the 12 months prior to Visit 1.
* Known or suspected contraindications to the study medications, including history of allergy to ACE-Inhibitors or ARBs.
* Upper arm circumference > 42 cm.
* Third shift or night workers.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 654
Dates: Start 2006-05; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Mean 24-hour ambulatory diastolic blood pressure (MADBP) change from baseline, after a missed dose, aliskiren 300 mg versus irbesartan 300mg.
from baseline.
Mean 24-hour ambulatory diastolic blood pressure (MADBP) change from baseline, after a missed dose, ramipril 10 mg versus irbesartan 300mg.

SECONDARY OUTCOMES:
efficacy on mean 24 hour ambulatory systolic blood pressure (MASBP) change
from baseline following a missed dose
efficacy on daytime and nighttime MASBP and MADBP change from baseline following a missed dose
efficacy on the MASBP and MADBP change from baseline following the last active dose prior to introducing a missed dose in any treatment group.
efficacy on the daytime and nighttime MASBP and MADBP change from baseline, following the last active dose prior to introducing a missed dose in any treatment group.
safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (2):
- Investigative Centers, Germany
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Result] Palatini P, Jung W, Shlyakhto E, Botha J, Bush C, Keefe DL. Maintenance of blood-pressure-lowering effect following a missed dose of aliskiren, irbesartan or ramipril: results of a randomized, double-blind study. J Hum Hypertens. 2010 Feb;24(2):93-103. doi: 10.1038/jhh.2009.38. Epub 2009 May 21. PMID 19458624